CLINICAL TRIAL: NCT03589989
Title: Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (The ESTxENDS Trial)
Brief Title: The ESTxENDS Trial- Electronic Nicotine Delivery Systems (ENDS/Vaporizer/E-cigarette) as an Aid for Smoking Cessation.
Acronym: ESTxENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); University of Zurich (Other); State Hospital, St. Gallen (Other Government); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332
Record Dates: First submitted 2018-06-19; First posted 2018-07-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ENDS (vaporizer/e-cig) and smoking cessation counseling
- Control group (Active Comparator)
  Interventions: Other: Smoking cessation counseling

INTERVENTIONS:
Other: ENDS (vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 6-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6 months, participants will be asked to come to a final clinical visit.
  Arms: Intervention group
Other: Smoking cessation counseling — Participants in the control group will receive smoking cessation counseling only. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 6-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6 months, participants will be asked to come to a final clinical visit.
  Arms: Control group

SUMMARY:
Cigarette smoking is the leading cause of preventable death in Switzerland and still more than a quarter of the Swiss population smokes cigarettes. Recently, electronic nicotine delivery systems (ENDS; also called vaporizer or electronic cigarette) have become popular with smokers who want to stop smoking or reduce their exposure to inhaled chemicals since ENDS use appears to be safer than tobacco smoking. Only two rigorous randomized controlled trials (RCTs) on the efficacy of ENDS to help smokers quit have been published so far. They have promising, yet inconclusive results, as the number of included participants were small. The safety and potential adverse effects of ENDS are also largely unknown. While the aerosol the users inhale appears safe in laboratory conditions, the difference in exposure to chemicals (such as reduction in exposure to volatile organic compounds) and effects of chemicals on the body (adverse events, improved health-related outcomes and measures of oxidative stress) between smokers who quit (with or without ENDS) and those who use ENDS for a long time have not yet been assessed in an RCT.

This study will therefore test the efficacy of ENDS for cigarette smoking cessation, the safety of ENDS on adverse events and the effect of ENDS on health-related outcomes and exposure to inhaled chemicals.

The primary hypothesis of this trial is that providing cigarette smokers willing to quit smoking tobacco cigarettes with ENDS leads to a higher rate of smokers who quit cigarette smoking than only smoking cessation counseling with nicotine replacement therapy (NRT), which represents nowadays the standard of care.

For this trial, cigarette smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants in the control group will receive smoking cessation counseling only. Participants in both groups will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 6-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date and again at week 1, 2, 4 and 8 after the target quit date. After 6 months, participants will be asked to come to a final clinical visit.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months,
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion Criteria:

* Known hypersensitivity or allergy to contents of the e-liquid
* Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the scheduled study intervention, i.e. within the first 6-months of the study
* Persons having used ENDS regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other medications with demonstrated efficacy as an aid for smoking cessation such as varenicline or bupropion within the 3 months preceding the baseline visit
* Persons who cannot attend the 6- month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Continuous smoking abstinence (1) | 6 months post quit date
  Self-report of having smoked no cigarettes from quit date, validated by urinary levels of anabasine. If anabasine is missing, validation by exhaled carbon monoxide (CO).

SECONDARY OUTCOMES:
Continuous smoking abstinence (2) | 6 months post quit date
  Self-report of having smoked no cigarettes from quit date, validated by urinary levels of NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol). If NNAL is missing, validation by urinary levels of anabasine or exhaled carbon monoxide (CO).
Self-reported smoking abstinence allowing a 2-week'grace period' | 4, 8 weeks and 6 months post quit date
  Smoking abstinence allowing a 2-week'grace period' after the target quit date.
Validated smoking abstinence allowing a 2-week'grace period' (1) | 6 months post quit date
  Smoking abstinence allowing a 2-week'grace period' after the target quit date, validated by urinary levels of anabasine. If anabasine is missing validation by exhaled carbon monoxide (CO).
Validated smoking abstinence allowing a 2-week'grace period' (2) | 6 months post quit date
  Smoking abstinence allowing a 2-week'grace period' after the target quit date, validated by urinary levels of NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol). If NNAL is missing, validation by urinary levels of anabasine or exhaled carbon monoxide (CO).
Self-reported smoking abstinence allowing up to 5 cigarettes | 1, 2, 4, 8 weeks and 6 months post quit date
  Smoking abstinence allowing up to 5 cigarettes in total after the target quit date.
Validated smoking abstinence allowing up to 5 cigarettes (1) | 6 months post quit date
  Smoking abstinence allowing up to 5 cigarettes in total after the target quit date, validated by urinary levels of anabasine. If anabasine is missing validation by exhaled carbon monoxide (CO).
Validated smoking abstinence allowing up to 5 cigarettes (2) | 6 months post quit date
  Smoking abstinence allowing up to 5 cigarettes in total after the target quit date, validated by urinary levels of NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol). If NNAL is missing, validation by urinary levels of anabasine or exhaled carbon monoxide (CO).
Self-reported 7-day point prevalence abstinence | 1, 2, 4, 8 weeks and 6 months post quit date
  Self-report of having smoked no cigarettes in the past seven days.
Validated 7-day point prevalence abstinence (1) | 6 months post quit date
  Confirmation of having smoked no cigarettes in the past seven days, validated by urinary levels of anabasine. If anabasine is missing validation by exhaled carbon monoxide (CO).
Validated 7-day point prevalence abstinence (2) | 6 months post quit date
  Confirmation of having smoked no cigarettes in the past seven days, validated by urinary levels of NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol). If NNAL is missing, validation by urinary levels of anabasine or exhaled carbon monoxide (CO).
Number of cigarettes smoked per day (CPD) | baseline, target quit date, 1, 2, 4, 8 weeks and 6 months post quit date
  self-reported
Change in number of cigarettes smoked per day (CPD) | baseline, 6 months post quit date
  self-reported. Successful reduction defined as 50% reduction in CPD.
Use of any other smoking cessation products (NRT, Nicotine replacement therapy) | 1, 2, 4, 8 weeks and 6 months post quit date
  self-reported on whether and how often they used any NRT.
Withdrawal | baseline and 6 months post quit date
  The physical signs and symptoms associated with withdrawal, measured using the Minnesota Tobacco Withdrawal Scale (http://www.med.uvm.edu/behaviorandhealth/minnwsdefault). The Minnesota Tobacco Withdrawal Scale measures self-reported severity of nicotine withdrawal. The measure has 15 items, with five possible responses (0-5), thus scores on the scale range from 0 to 60.
Nicotine dependence | baseline and 6 months post quit date
  Nicotine dependence measured using the Fagerström Test. The Fagerström Test for Nicotine Dependence (FTND, Heatherton TF et al., 1991) is a standard instrument for assessing the intensity of physical addiction to nicotine. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. Two items have four possible responses (0-3) and four items have two possible responses (0-1). The nicotine dependence score ranges from 0 to 10. A score between 0 and 2 is considered as a low nicotine dependence, a score between 3 to 5 is considered as a medium nicotine dependence, a score between 6 and 7 is considered as a high nicotine dependence and a score between 8 and 10 is considered as a very high nicotine dependence.
Health-related quality of life | baseline and 6 months post quit date
  Measured using the Swiss EQ-5D. The EQ-5D questionnaire is a standardized measure of health status developed by the EuroQol Group (https://euroqol.org/). EQ-5D questionnaires have five dimensions: "Mobility", "Self-care," "Usual Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by five problem levels corresponding to participant response choices.
Use of any ENDS | 1, 2, 4, 8 weeks and 6 months post quit date
  self-reported on whether and how often they used any ENDS
Report on most common adverse events using ENDS | 1, 2, 4, 8 weeks and 6 months post quit date
  Any unfavorable and unintended sign, symptom, or disease temporally associated with the use of ENDS, whether or not it is considered related to the product.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med, Study Director — Berner Institut für Hausarztmedizin; Universität Bern
Locations (5):
- Switzerland (5):
  - Unisanté, Centre universitaire de médecine générale et santé publique, Université de Lausanne, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Département de médecine interne, Hôpitaux universitaires de Genève, Geneva
  - Lungenzentrum, Klinik für Pneumologie und Schlafmedizin, Kantonsspital St. Gallen, Sankt Gallen
  - Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich

REFERENCES:
- [Background] Bullen C, Howe C, Laugesen M, McRobbie H, Parag V, Williman J, Walker N. Electronic cigarettes for smoking cessation: a randomised controlled trial. Lancet. 2013 Nov 16;382(9905):1629-37. doi: 10.1016/S0140-6736(13)61842-5. Epub 2013 Sep 9. PMID 24029165
- [Background] Caponnetto P, Campagna D, Cibella F, Morjaria JB, Caruso M, Russo C, Polosa R. EffiCiency and Safety of an eLectronic cigAreTte (ECLAT) as tobacco cigarettes substitute: a prospective 12-month randomized control design study. PLoS One. 2013 Jun 24;8(6):e66317. doi: 10.1371/journal.pone.0066317. Print 2013. PMID 23826093
- [Background] Hartmann-Boyce J, McRobbie H, Bullen C, Begh R, Stead LF, Hajek P. Electronic cigarettes for smoking cessation. Cochrane Database Syst Rev. 2016 Sep 14;9(9):CD010216. doi: 10.1002/14651858.CD010216.pub3. PMID 27622384
- [Background] Malas M, van der Tempel J, Schwartz R, Minichiello A, Lightfoot C, Noormohamed A, Andrews J, Zawertailo L, Ferrence R. Electronic Cigarettes for Smoking Cessation: A Systematic Review. Nicotine Tob Res. 2016 Oct;18(10):1926-1936. doi: 10.1093/ntr/ntw119. Epub 2016 Apr 25. PMID 27113014
- [Background] Farsalinos KE, Polosa R. Safety evaluation and risk assessment of electronic cigarettes as tobacco cigarette substitutes: a systematic review. Ther Adv Drug Saf. 2014 Apr;5(2):67-86. doi: 10.1177/2042098614524430. PMID 25083263
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Derived] Auer R, Schoeni A, Humair JP, Jacot-Sadowski I, Berlin I, Stuber MJ, Haller ML, Tango RC, Frei A, Strassmann A, Bruggmann P, Baty F, Brutsche M, Tal K, Baggio S, Jakob J, Sambiagio N, Hopf NB, Feller M, Rodondi N, Berthet A. Electronic Nicotine-Delivery Systems for Smoking Cessation. N Engl J Med. 2024 Feb 15;390(7):601-610. doi: 10.1056/NEJMoa2308815. PMID 38354139
- [Derived] Nyilas S, Bauman G, Korten I, Pusterla O, Singer F, Ith M, Groen C, Schoeni A, Heverhagen JT, Christe A, Rodondi N, Bieri O, Geiser T, Auer R, Funke-Chambour M, Ebner L. MRI Shows Lung Perfusion Changes after Vaping and Smoking. Radiology. 2022 Jul;304(1):195-204. doi: 10.1148/radiol.211327. Epub 2022 Apr 5. PMID 35380498